CLINICAL TRIAL: NCT06396923
Title: The Effect of Listening to Music on Anaerobic Power in Elite Weightlifting Athletes
Brief Title: The Effect of Music on Weight Lifters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: karataylifting
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-04

CONDITIONS: Exercise Overtraining
MeSH Terms: conditions — Overtraining Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): Participants will complete a series of 3 x 15-second repeated Wingate Anaerobic Tests (WAnTs) on an electronically braked bicycle ergometer. Participants will warm up for 5 minutes at a no-load resistance. Resistance to the test will be calculated using 7.5% of the participant's body mass. Upon successful completion of each WAnT, performance variables, heart rate, rate of perceived exertion (RPE; Scale 1-10), and motivation rating will be obtained. Motivation will be achieved using a visual analogue scale with a 100 mm line. Participants will indicate how motivated they were to exercise during WAnT, from most motivated ever to least motivated. Scores will be obtained by measuring from zero to the point marked on the 100 mm line. All anaerobic performance measurements will be calculated during each 15-second WAnT period via Velotron Software (v4 1.0.6 Velotron, Racermate Inc., Seattle, WA, USA).
  Interventions: Diagnostic Test: Wingate test
- Music group (Experimental): The same exercise protocol will be applied. However, participants in the music group will complete the test by listening to the music of their own choosing. (The same headphones will be used to play music with the same electronic device, and the device will be set to the same volume for all participants.)
  Interventions: Diagnostic Test: Wingate test

INTERVENTIONS:
Diagnostic Test: Wingate test — Wingate Anaerobic Power Test is based on maximal pedaling on a bicycle ergometer against a predetermined constant load to provide the highest mechanical power for 30 seconds. During the test, measurements are made automatically at intervals of five seconds and six equal intervals. As a result of these measurements, some data are obtained that allow us to obtain information about anaerobic performance.

SUMMARY:
The effects of listening to music on anaerobic power in elite weightlifting athletes will be examined.

DETAILED DESCRIPTION:
The aim of the study was to investigate the effects of music listening on anaerobic power in elite weightlifting athletes.There is no study in the literature examining the relationship between music listening and anaerobic power in elite weightlifting athletes. Since our study will be the first to investigate the subject, we foresee that it is scientifically important and will shed light on future studies. In addition, national or international publications are planned after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Being an elite weightlifter, volunteering for research

Exclusion Criteria:

* If you have any disability that may prevent the test, hearing problems

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Wingate anaerobic power test | baseline
  Peak Power (Maximum Anaerobic Power): The highest mechanical power achieved in any five-second period during the test.
  Average Power (Maximum Anaerobic Capacity): It is the average power generated during the test.
  Lowest Power (Minimum Power): The lowest mechanical power achieved during any five-second period during the test.
  Fatigue Index: It expresses the decrease in strength that occurs during the test as a percentage. It is calculated by dividing the difference between the highest power value and the lowest value obtained within any five-second period during the test by the highest power value obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Savaş Torlak, Karatay, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No